CLINICAL TRIAL: NCT06271694
Title: Impairments and Personal Factors Associated With Activity and Participation in Vestibular Rehabilitation
Brief Title: Activity and Participation in Vestibular Disorders
Acronym: APV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Brooke Klatt, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY22020027; 1K23DC020215-01 (NIH)
Record Dates: First submitted 2024-01-11; First posted 2024-02-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Vestibular Disorder
Keywords: Vestibular Rehabilitation; Activity and Participation
MeSH Terms: conditions — Vestibular Diseases; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard Vestibular Rehabilitation (Other): All participants will receive standard vestibular rehabilitation
  Interventions: Other: Vestibular Rehabilitation

INTERVENTIONS:
Other: Vestibular Rehabilitation — Standard vestibular rehabilitation

SUMMARY:
This study will examine whether impairments and personal factors are associated with activity and participation in people with vestibulopathy. Data collection will occur prior to starting vestibular rehabilitation and after completing vestibular rehabilitation.

DETAILED DESCRIPTION:
Adults aged 18-years and older with symptomatic complaints of dizziness and/or imbalance and a medical diagnosis of unilateral vestibular hypofunction will be recruited at the time of their entry into vestibular rehabilitation. The investigators will analyze what factors (impairments and personal factors) are related to activity and participation in people with vestibular disorders and see if change in activity and participation is related to recovery from vestibulopathy.

ELIGIBILITY:
Inclusion Criteria:

- 18-years and older with symptomatic complaints of dizziness and/or imbalance and a medical diagnosis of unilateral vestibular hypofunction

Exclusion Criteria:

* 1. Cognition <18 on Montreal Cognitive Assessment (MoCA)
* 2. Visual acuity worse than 20/40 with corrected lenses
* 3. Loss of protective distal sensation (defined as the inability to feel a 4.31 size monofilament on the plantar surface of the foot)
* 4. Inability to engage in community mobility

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Late-life Function and Disability Instrument | 8-weeks
  Activity and Participation (raw 16-80; scale 0-100 min-max scores); higher is better
Dizziness Handicap Inventory | 8-weeks
  Dizziness disability; 0-100 (min-max score); higher is greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Klatt, PhD, Principal Investigator — Assistant Professor
Locations (1):
- UPMC-Rehab Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data that underlie the results reported in the article could be shared with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following article publication. No end date.
Access Criteria: To gain access to data requestors will need to sign a data access agreement and proposals should be directed at klattresearch@pitt.edu